# A Comparative Study between Dissociative Treatment and Binocular Interactive Treatment in Amblyopia

#### **Thesis**

Submitted to Faculty of Medicine – Ain Shams University
In Partial Fulfillment of the Requirements of Doctorate Degree in Ophthalmology
By

#### Suha Ahmed Amin Moustafa Hussein

M.B,B.C.h (2009), M.Sc (2014),

Faculty of medicine - Ain Shams University

Under supervision of

# Professor Dr. Hazem Hosny Nouh

Professor of Ophthalmology Faculty of medicine – Ain Shams University

#### Professor Dr. Mohammad Ahmad Rashad

Professor of Ophthalmology Faculty of medicine – Ain Shams University

# Dr. Walid Mohamed Abd El-Raouf El-Zawahry

Lecturer of Ophthalmology
Faculty of medicine – Ain Shams University

### Dr. Ahmad Taha Ismail

Lecturer of Ophthalmology Faculty of medicine – Ain Shams University

> Faculty of medicine Ain Shams University Cairo – Egypt 2022

## STATISTICAL ANALYSIS PLAN

Using the SPSS (or the Minitab or Mega Stat) statistical software, the data will be examined using standard summary statistics which will include, where appropriate, 95% confidence intervals.

A one-way analysis of variance (ANOVA) will be performed on the visual acuity data to determine whether there appeared to be an effect of measurement time on visual acuity, and pairwise comparisons of mean will then be performed, examing the changes from baseline to 1 month, 3 months and 6 months after treatment start.

An improvement of  $\geq 0.125$  LogMAR units will be considered clinically significant. In addition, the proportion of change will be calculated at 1 month, 3 months and 6 months follow up as follows (using the formula described by Stweart et al)

Proportion of change =  $VA_{as} - VA_{ae} / VA_{as} - VA_{fe}$ 

Where  $VA_{as}$  is the vision of amblyopic eye at baseline,  $VA_{ae}$  is the vision of amblyopic eye at the end of the treatment (i.e. 6months) and  $VA_{fe}$  is the vision of the non-amblyopic eye at the end of the treatment.

Also percentage of compliance with treatment in each group will be measured as a secondary outcome measure.